CLINICAL TRIAL: NCT00000214
Title: IV Cocaine Abuse: A Laboratory Model
Brief Title: IV Cocaine Abuse: A Laboratory Model - 3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Columbia University (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NIDA-06234-3; R01DA006234 (NIH); R01-06234-3
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2012-12

CONDITIONS: Cocaine-Related Disorders
Keywords: intravenous abuse
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to evaluate the effects of buprenorpine on cocaine taking and on the physiological and subjective effects of cocaine, including cocaine craving in non-opiate dependent cocaine users.

ELIGIBILITY:
Please contact site for information.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1992-01; Primary Completion 1993-01 (Actual); Study Completion 1993-01 (Actual)

PRIMARY OUTCOMES:
Direct cocaine effects (caridio, subjective)
Interaction of coc/bup on cardio measures
Ineraction of coc/bup on coc's subjective effects
Effects of buprenorphine on cocaine craving

CONTACTS AND LOCATIONS:
Overall Officials: Richard Foltin, Ph.D., Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

REFERENCES:
- [Background] Behav Pharm 1994, vol 5: 79-89